CLINICAL TRIAL: NCT06363266
Title: A SMART Design to Optimize the Delivery of TEMPO - a Tailored, wEb-based Psychosocial and Physical Activity Self-Management PrOgram for Men With Prostate Cancer and Their Caregivers
Brief Title: A SMART Design to Optimize the Delivery of TEMPO for Men With Prostate Cancer and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's Research Center, Canada (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); University of Calgary (Other); Sunnybrook Health Sciences Centre (Other); University of British Columbia (Other); McGill University (Other); Simon Fraser University (Other); Université de Sherbrooke (Other); Memorial University of Newfoundland (Other); Université de Montréal (Other); CISSS de Laval (Unknown)
Responsible Party: Principal Investigator, Sylvie Lambert, Associate Professor, St. Mary's Research Center, Canada
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: MP-18-2025-1156
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Cancer of the Prostate; Anxiety
Keywords: Behavior Change; Caregivers; Coping; E-Health; Illness Self-Management; Physical Activity; Psychosocial Oncology; Self-Directed Interventions; Web-Based Interventions
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders; Motor Activity | interventions — TEMPO

STUDY DESIGN:
Intervention Model Description: Using a stepped care approach, TEMPO will be provided across two intervention stages with variations on timing (initial vs. delayed) and intensity (self-directed vs. guided). All dyads will continue to access usual care (a co-intervention measure is included).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TEMPO (Experimental): Using a stepped care approach, TEMPO will be provided across two intervention stages with variations on timing (initial vs. delayed) and intensity (self-directed vs. guided). All dyads will continue to access usual care (a co-intervention measure is included).
  Interventions: Behavioral: TEMPO
- Actively Monitoring dyads' anxiety (Active Comparator): Patients will receive usual care throughout the study.
  Interventions: Other: Active Monitoring dyads' anxiety

INTERVENTIONS:
Behavioral: TEMPO — Stage 1 interventions (weeks 1-12): TEMPO.
  After 12 weeks, the benefit of the initial assignment will be assessed. Benefit is defined as a score < 3 on the ESAS-r anxiety item (range 0-10) or a decrease >= 2 points from eligibility screening. If both dyad members had anxiety symptoms at recruitment, both must meet the benefit criterion. If one member no longer meets the criterion, the dyad is considered "did not benefit."
  Stage 2 interventions (weeks 13-25): TEMPO or lay guidance.
  1. TEMPO responders will continue with TEMPO. Dyads who did not benefit will be re-randomized to:
     1. Stepping up to lay guidance (8 x 20-minute calls via phone or Teams). Guides will receive TEMPO training and conduct semi-structured exit interviews.
     2. More time with TEMPO for dyads who benefited from it.
  2. Non-responders to usual care in Stage 1 will be stepped up to TEMPO.
  Other Names: Tailored, wEb-based, Psychosocial and Physical Activity Self- Management PrOgramme
  Arms: TEMPO
Other: Active Monitoring dyads' anxiety — Stage 1 interventions (week 1-12): Patients will receive usual care throughout the study. Dyads in this group will not receive any information resources from the research team but will have access to all of those available at their participating center (sites will be asked to provide a description of usual care practices).
  Stage 2 interventions (week 13-25): Dyads not responding to active monitoring will be stepped up to TEMPO; responders to active monitoring will only be invited to complete the follow-up measures.
  Arms: Actively Monitoring dyads' anxiety

SUMMARY:
Men with prostate cancer and their family caregivers face many physical and emotional challenges from the cancer itself and its treatment(s), which often lead to high anxiety. The pandemic has highlighted the importance of protecting our physical and mental health, and the complex responsibilities that caregivers have in supporting their loved ones. To improve the health of men with prostate cancer and of their caregivers, the research team developed TEMPO: a self-directed Tailored, wEb-based, psychosocial and physical activity self-Management PrOgram. TEMPO was developed with men with prostate cancer and their caregivers over the past 8 years. It also combines the investigators' research conducted over the past decade on providing the best support to those affected by cancer. Because the cancer care workforce is already overstretched, the research team designed TEMPO to be used without guidance from a health care professional. TEMPO is one-of-a kind in its support of both patients and caregivers, and the integration of coping skills training on a wide range of cancer challenges along with a home-based exercise program. Patients and caregivers who have used TEMPO said they improved their communication, learned new skills to cope with both physical and emotional challenges of cancer, and increased their physical activity. The present project builds on this work to further evaluate the cost and impact of TEMPO on men's and caregivers' health. Men with prostate cancer and their caregivers will be assigned by chance to one of two groups a) TEMPO or b) monitor their anxiety for 12 weeks. After 12 weeks, patients' and caregivers' needing more support will be identified based on an assessment of their anxiety level. For those already using TEMPO and needing more support, non-health care professional guidance might be offered. All those in the monitoring group needing more support will now have access to TEMPO. All participants complete surveys to determine whether TEMPO led to improved health outcomes.

DETAILED DESCRIPTION:
BACKGROUND : Up to 60% of men with prostate cancer report some level of anxiety, with clinical levels exceeding population norm. Anxiety results from reactions to the diagnosis, treatment side effects, and the multitude of other anxiety-provoking physical and psychosocial challenges (e.g., treatment decision-making) men face daily. These challenges can be successfully mitigated through self-management, defined as one's actions and decisions to confidently manage medical aspects of cancer, cope with emotions, adjust everyday life, and enhance recovery (e.g., via lifestyle changes). Cancer care lags in the implementation of self-management support, mostly because it requires clinicians' engagement, which conflicts with their limited availability, even if self-management is cost-effective. Men then often lack knowledge for effective self-management; cancer challenges often persist, along with the anxiety they provoke. Cancer challenges are not self-managed in a vacuum; family caregivers are often relied on. The impact of caregiving is substantial, but often dismissed, resulting in high caregiver anxiety. TEMPO, a self-directed, dyadic Tailored, wEb-based psychosocial and physical activity self-Management PrOgram, was developed because staff shortages necessitate innovative models to deliver sustainable self-management support, without compromising efficacy. TEMPO is a tool to help address the quadruple aim of healthcare: enhance dyads' and clinicians' experiences and improve health outcomes at low cost. However, in a pilot study, some dyads needed more guidance to use TEMPO. Barriers to use were mostly motivational, which the investigators previously found can be effectively addressed by guidance from non-health care professionals to spare clinical resources.

OBJECTIVES : The goal of this study is to determine the most efficacious and cost-effective way of adapting TEMPO to dyads' needs for guidance. The primary hypotheses are that a) TEMPO dyads will experience lower anxiety than active monitoring dyads, but dyads needing guidance will report lower anxiety post guided TEMPO than if they had continued with TEMPO self-directed; and b) TEMPO will be cost-effective compared to active monitoring; adding guidance will demonstrate cost-effectiveness among those needing it. For the secondary hypotheses, same effects are expected of TEMPO and guidance on the secondary outcomes and between-group differences in anxiety will be higher among caregivers who are mostly females and women.

METHODOLOGY : This multicenter study is a stratified Sequential Multiple Assignment Randomized Trial (SMART) across Canada with two sequential intervention stages, cost-effectiveness analysis, and exit qualitative interviews. Study activities will be coordinated out of St Mary's Research Centre in Montreal. Using a stepped care approach, TEMPO will be provided across two intervention stages with variations on timing (initial vs. delayed) and intensity (self-directed vs. guided). At each centre, clinical collaborators (physicians, nurses, trial nurse, secretaries etc) may provide brief information on the study to the target population before, during or after an appointment. At this time, interested individuals may be given a study pamphlet or be directed to a displayed poster and the clinical collaborator will obtain permission for a RA to approach them. Further recruitment strategies may include: direct approaches of patients by the RA in the waiting room; invitation letters sent to all patients in the target population matching certain key inclusion criteria without specifically singling out any individual patients including RA contact information; advertisement of the study on social media including contact information of the research team; contact by email of individuals within the target population who have been identified by the investigators during previous research activities.

Depending on the way interested individuals were identified, the RA will use the content of the consent form and the study pamphlet to explain the study in detail. All screening will be done as a structured interview in-person or over the phone where the RA will complete the eligibility form with patients and their caregivers. The form might be sent to potential participants directly to complete online. If the caregiver is not present, the RA will provide study information to the patient and obtain his/her verbal consent to follow-up by phone within the next week to determine the caregiver's interest in the study. In addition, each site will display study posters giving potential participants the ability to self-refer.

Eligible patients and caregivers will be issued a consent form in their preferred format, depending on the recruitment context. Once the consent form is received, the link to the online baseline (T0) questionnaire will be emailed. Patient-caregiver dyads returning their consent forms and baseline questionnaires (T0) will be initially randomized by the study coordinator to either a) TEMPO self-directed or b) active monitoring of anxiety. After 12 weeks, TEMPO dyads still reporting anxiety will be re-randomized to more time with TEMPO or TEMPO plus guidance, and active monitoring dyads will be offered TEMPO. All participating dyads will continue to access usual care (a co-intervention measure is included). Group allocation will not be blinded. Dyads will be blinded to hypotheses to reduce bias. Research assistants (RAs) will not interact with randomized participants until the exit interview. Guides are not therapists; they focus on adherence, using TEMPO to answer dyads' questions. Phone calls start with the guide and dyad setting an agenda. Guides then ask about TEMPO's use since the last call. Guides conclude calls by reviewing dyad's goals until the next call. Stages 1 and 2 are 12 weeks each. Outcomes are assessed prior to randomization (baseline, T0) and at completion of Stage 1 (11 weeks post-randomization, T1) and Stage 2 (22 weeks post-randomization, T2).

SIGNIFICANCE :This proposal builds on the investigators' innovative work on efficient, evidence-based dyadic self-management interventions that spare clinical resources but remains efficacious. Clinician partners emphasize the value of TEMPO in their letters of support. Twice as many centres are participating in this trial, compared to the pilot. The research team will make cost-effectiveness recommendations with clinical implementation in mind. Importantly, TEMPO has significant generalizability, as the tools and approaches can readily be adapted to other cancer populations (see letter from Stuart Edmond, Canadian Cancer Society). TEMPO is currently being adapted for use among patients with a head and neck cancer and their caregivers for implementation at the Hospital Center of the University of Montreal. Several Cancer Agencies are exploring TEMPO's integration in their resource infrastructure. However, a definitive trial on efficacy, cost-effectiveness, and adaptation to meet dyad's needs for guidance is needed. The research team will also contribute to the emerging literature on SMARTs for behavioral interventions.

ELIGIBILITY:
Patient inclusion criteria: Prostate cancer diagnosis; Treatment for prostate cancer (excluding active surveillance) scheduled to start or received within the past 2 years; Nominate a caregiver willing to participate; Report at least moderate anxiety (ESAS-r Anxiety 3+); Be able to read English or French; Have access to the internet

Caregiver inclusion criteria: Are nominated by patient as primary support person; Are patients' spouse, partner, or other family member; If patient does not report moderate anxiety, caregiver needs to; Be able to read English or French; Have access to the internet

Exclusion criteria for patient and caregiver: Hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | T0: Baseline; T1: 13 weeks post-baseline; T2: 25 weeks post-baseline
  The primary outcome is anxiety to compare TEMPO vs. usual care at 13 weeks and within the TEMPO group, the impact of re-randomizing those who do not benefit from TEMPO to 1a) TEMPO + lay guidance vs. 1b) continue with TEMPO at 25 weeks. The primary measure will be the 7-item Hospital Anxiety and Depression Scale (HADS) - Anxiety subscale, which was used in the research teams' pilot and has strong and validity to assess anxiety symptoms among dyads, including responsiveness. A psychometric review of anxiety and depression questionnaires used with patients with cancer identified the HADS as one of the questionnaires with the strongest psychometric properties. The scale range is 0-21. Subscale scores of 0-7 are categorized as normal, subscale scores of 8 to 10 are categorized as borderline and scores of 11 to 21 as clinical anxiety.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | T0: Baseline; T1: 13 weeks post-baseline; T2: 25 weeks post-baseline
  10 items that measure the degree participants appraise situations in their life as stressful. Each question rated on a 5-point Likert scale, and a summary score obtained by summing all 10 items. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress, scores ranging from 14-26 would be considered moderate stress, and scores ranging from 27-40 would be considered high perceived stress.
Patient-Reported Outcome Measurement Information System (PROMIS) Self-Efficacy Scale | T0: Baseline; T1: 13 weeks post-baseline; T2: 25 weeks post-baseline
  4 items measuring self-efficacy to manage difficult situations and find solutions. Raw scores range from 4-20. Higher scores indicate higher perceived general self-efficacy, lower scores indicate lower perceived general self-efficacy.
Health Education Impact Questionnaire (heiQ) | T0: Baseline; T1: 13 weeks post-baseline; T2: 25 weeks post-baseline
  The Health Education Impact Questionnaire (heiQ) includes eight independent dimensions to measure self-management strategies. Given the aim of TEMPO six of the eight dimensions will be given: (a) positive and active engagement in life, (b) skill and technique acquisition, (c) constructive attitude and approaches, (d) self-monitoring and insight, (e) health services navigation, and (f) social integration and support.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | T0: Baseline; T1: 13 weeks post-baseline; T2: 25 weeks post-baseline
  Participants are asked to indicate: "How many times per week on average did you do the following kinds of exercise over the past month?" The following kinds of exercise include: mild, moderate and strenuous.
Dyadic Coping Inventory (DCI) | T0: Baseline; T1: 13 weeks post-baseline; T2: 25 weeks post-baseline
  37 items to capture how partners support one another in response to stressors. Items are rated on a 5-point scale from 1 = very rarely to 5= very often
SF-12 | T0: Baseline; T1: 13 weeks post-baseline; T2: 25 weeks post-baseline
  The 12-item Short Form Health Survey (SF-12)99 measures quality of life, and includes a physical component score (PCS) and a mental component score (MSC). Scores are standardized from 0-100
Hospital Anxiety and Depression Scale (HADS) depression subscale | T0: Baseline; T1: 13 weeks post-baseline; T2: 25 weeks post-baseline
  The 14 items on the Hospital Anxiety and Depression Scale (HADS) are equally divided between the HADS-Anxiety and HADS-Depression subscales. The scale range is 0-21. Subscale scores of 0-7 are categorized as normal, subscale scores of 8 to 10 are categorized as borderline and scores of 11 to 21 as clinical depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Lambert, PhD, Principal Investigator — McGill University
Locations (2):
- Canada (2):
  - St Mary's Hospital Research Centre, Montreal, Canada
  - St. Mary's Research Centre, Montreal, Quebec